CLINICAL TRIAL: NCT03330418
Title: A Phase III Study of RC18, a Recombinant Human B Lymphocyte Stimulator Receptor:Immunoglobulin G( IgG ) Fc Fusion Protein for Injection for the Treatment of Subjects With Neuromyelitis Optica Spectrum Disorders.
Brief Title: A Phase III Study of TACI-antibody Fusion Protein Injection (RC18) in Subjects With Neuromyelitis Optica Spectrum Disorders
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C009NMOSDCLLI
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica | interventions — RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Experimental): Participants received placebo weekly administered subcutaneously for 48 times in the double-blind treatment period.Once the participants relapse,they should advance to the open phase.All participants were treated with the test drugs.
  Interventions: Biological: Placebo
- RC18 160 mg (Experimental): Patients received the test group RC18 160mg weekly administered subcutaneously for 48 times.Starting with the forty-ninth dose,the trial went into the open phase . All participants were treated with the test drugs.
  Interventions: Biological: RC18 160 mg

INTERVENTIONS:
Biological: Placebo — Starting with the forty-ninth dose,the trial went into the open phase. All participants were treated with the test drugs.
  Arms: Placebo Comparator
Biological: RC18 160 mg — In the Phase B,the researchers can adjust the dose of RC18 according to the subjects' willingness and recurrence, but the maximum dose of single dose should not exceed 320g.
  Arms: RC18 160 mg

SUMMARY:
The purpose of this study is to initially observe the safety and effectivity of RC18 in Participants with Neuromyelitis Optica Spectrum Disorders.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 2015 international consensus diagnostic criteria for Neuromyelitis Optica Spectrum Disorders and astrocyte water channel aquaporin-4 (AQP4) antibody positivity.
* EDSS 0-7.5
* Clinical evidence of at least 2 relapses within the first two years of randomization and/ or 1 relapse within the first one year of randomization
* Consent to use effective contraception during the study period (women of childbearing age)
* Voluntarily signed informed consent

Exclusion Criteria:

* Abnormal laboratory parameters need to be excluded, including but not limited to:
* Currently suffering from active hepatitis or serious liver disease and medical history
* Patients were treated with rituximab or other monoclonal antibodies within 6 months prior to randomization .
* Any concomitant disease other than neuromyelitis optica（NMO）/ neuromyelitis optica Spectrum disorders（NMOSD）that required treatment with lucocorticoid.
* pregnant , lactating women and men or women who have birth plans during the research;
* Have a history of allergic reaction to contrast agent for parenteral administration and human biological medicines.
* Receipt of intravenous immune globulin （ IVIG） within 28 days prior to randomization.
* Receipt of any of the following prior to randomization: Azathioprine,Cyclosporin, Methotrexate Mitoxantrone,Cyclophosphamide,Tocilizumab,Tacrolimus,Mycophenolate,and Patients discontinued more than 5 times the half-life of the drug before they could get into the group .If the patients taking leflunomide and teriflunomide,they should need to take colestyramine for elution.
* Have participated in any clinical trial in the first 28 days of the initial screening or 5 times half-life period of the study compound (taking shorter time ).
* The patients have severe psychiatric symptoms and are not compatible with clinical studies
* Malignant tumor patients ;
* patients experienced any of the following events within 12 weeks before screening : myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association class IV heart failure
* Patients can't accept magnetic resonance imaging inspection during the trial.
* Infection with herpes zoster or HIV virus at the screening;
* The anti-hepatitis C virus （anti-HCV） of patients show positive;
* Investigator considers candidates not appropriating for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to first relapse after randomization | 144 weeks

SECONDARY OUTCOMES:
Change from Baseline in Expanded Disability Status Scale (EDSS) Score at week 4,8,12,24,36,48,60,72,96,120,144 | 144 weeks
  The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death) in half-point increments.
Change from Baseline in Hauser Ambulation Index at week 4,8,12,24,36,48,60,72,96,120,144 | week 4,8,12,24,36,48,60,72,96,120,144

CONTACTS AND LOCATIONS:
Overall Officials: xianhao Xu, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China